CLINICAL TRIAL: NCT07402590
Title: Randomized, Double-Blind, Placebo-Controlled Investigation to Validate the Efficacy and Safety of an Auditory Stimulation Treatment During Sleep to Improve Cognitive Abilities Related to Long-Term Memory in Amnestic Mild Cognitive Impairment (aMCI)
Brief Title: Auditory Stimulation During Sleep to Enhance Long-Term Memory in Amnestic MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitbrain (Industry)
Collaborators: Hospital Miguel Servet (Other); Hospital Clínico Universitario Lozano Blesa (Other); Hospital Royo Villanova de Zaragoza (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P-4-AS; C.I PI24/517 (Other: Comité de Ética de la Inv. de la Comunidad Autónoma de Aragón)
Record Dates: First submitted 2025-03-17; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mild Cognitive Impairment (MCI); Amnestic Mild Cognitive Impairment - aMCI; Alzheimer or Mild Cognitive Impairment
Keywords: MCI; auditory stimulation; amnestic mild cognitive impairment (aMCI); sleep; memory consolidation; alzheimer disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Acoustic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auditory stimulation first (Other): This arm receives auditory stimulation in the first experimental night ("Night 1") and placebo stimulation in the second night ("Night 2").
  Interventions: Procedure: Auditory Stimulation; Procedure: Placebo stimulation
- Placebo stimulation first (Other): This arm receives placebo stimulation in the first experimental night ("Night 1") and auditory stimulation in the second night ("Night 2").
  Interventions: Procedure: Auditory Stimulation; Procedure: Placebo stimulation

INTERVENTIONS:
Procedure: Auditory Stimulation — Brief auditory stimuli (50-ms bursts of pink noise) are delivered to patients once they have entered stable non-rapid eye movement (NonREM) sleep. The volume is automatically adjusted to optimize the induction of targeted neural oscillations, specifically slow waves and sleep spindles, while minimizing the risk of arousal.
  Other Names: Elevvo Audistim
Procedure: Placebo stimulation — All procedures are identical to the Auditory stimulation condition but the tone volume is set to 0.

SUMMARY:
This study aims to evaluate the efficacy and safety of Elevvo AudiStim, a sleep auditory stimulation device, as a symptomatic treatment for patients with amnestic mild cognitive impairment (aMCI).

DETAILED DESCRIPTION:
Amnestic Mild Cognitive Impairment (aMCI) is a precursor of dementia that involves memory impairment as a primary symptom. The condition presents a valuable opportunity for intervention before a potential progression to more severe, life-altering stages. A technique called "auditory stimulation during sleep" has previously been shown to improve memory by triggering neural oscillations such as slow waves and sleep spindles, which are implicated in memory processing. We hypothesize that the technique might improve memory also in patients with aMCI. This investigation is thus designed to systematically assess both the product's efficacy as a symptomatic treatment for patients with amnestic mild cognitive impairment (aMCI) and its overall safety profile.

After an initial calibration night ("Night 0"), two experimental nights will be performed ("Night 1" and "Night 2"), separated by 14 days. 7 days after each experimental night, a daytime long-term follow-up will be performed ("LT1" and "LT2"). Participants will receive either real or sham auditory stimulation during sleep, such that all participants will participate in both these conditions in a randomized balanced order.

ELIGIBILITY:
Inclusion Criteria:

* Age range > 50 years and ≤ 75 years
* Native Spanish speaker
* Normal or corrected-to-normal color vision
* Diagnosis of Alzheimer's disease with an amnestic phenotype at the mild cognitive impairment stage, confirmed according to the current clinical criteria of NIA-AA (2024) and IWG (2024), as well as the clinical protocols of the treating hospital
* Sufficient hearing without the use of a hearing aid (participant with a hearing threshold of 50 dB or higher in the calibration night hearing test will be excluded)

Exclusion Criteria:

* Patients with severe and/or complex chronic systemic diseases: Advanced heart disease, Advanced chronic kidney disease, for example, stage 4 or 5, Severe lung disease, such as GOLD stage III-IV COPD, Metastatic or end-stage cancer, Severe hematologic disorders, Active or chronic uncontrolled infectious diseases (e.g., untreated HIV)
* Evidence of strategic infarcts or other findings on neuroimaging that could be the cause of secondary cognitive impairment
* Abuse of alcohol or other psychotropic substances
* Diagnosed for depression or any severe psychiatric disorder in the 5 years prior to the evaluation
* Changes in treatment with benzodiazepines or antidepressants in the 6 months prior to the initial evaluation
* Treatment with neuroleptics
* Epilepsy with active treatment (within the last 5 years) or any comorbidity with a neurological disease that may cause cognitive impairment or brain damage
* Illiteracy
* Moderate or severe sleep apnea (without CPAP during the study)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Performance (pre vs post-sleep) in a word pair association task | Immediate recall: right before Nights 1/2 (1 hour before going to sleep); Morning recall: right after Nights 1/2 (1 hour after waking up); Long-term recall: during LT 1/2 (7 days after the start day of Nights 1/2).
  Memory performance in this task is measured as the number of word pairs recalled during morning and long-term recall, subtracted from the number of word pairs indicated during immediate recall. This metric will be compared between the two experimental conditions.
Performance (pre vs post-sleep) in a visuospatial memory task | Immediate recall: right before Nights 1/2 (1 hour before going to sleep); Morning recall: right after Nights 1/2 (1 hour after waking up); Long-term recall: during LT 1/2 (7 days after the start day of Nights 1/2).
  Memory performance is measured as the number of recognized images and correctly indicated image locations during morning and long-term recall, subtracted from the respective numbers during immediate recall. This metric will be compared between the two experimental conditions.

SECONDARY OUTCOMES:
Working memory performance | Morning recall: right after Nights 1/2 (1 hour after waking up); Long-term recall: during LT 1/2 (7 days after the start day of Nights 1/2).
  Working memory performance will be measured by the number of correct responses in the Sternberg task, administered after sleep in both conditions. This metric will be compared between conditions to evaluate the effect of the intervention.
Slow wave and sleep spindle activity | Throughout Nights 1/2.
  Neural oscillations will be analyzed using event detection to estimate event rates (incidences per minute) and event amplitudes (uV), as well as spectral analysis to quantify power (uV2/Hz) across relevant frequencies. The results will be evaluated by calculating linear correlations between these metrics (sleep spindle rate, amplitude, power, as well as slow-wave rate, amplitude, and power) and the two primary endpoints.
Sleep macrostructure - Total Sleep Time | Throughout Nights 1/2.
  Sleep macrostructure will be measured using the scoring manual of the American Academy of Sleep Medicine (AASM; Iber et al., 2007) as the established standard. Obtaining the sleep stage for each 30-sec epoch of the recording, allows the total sleep time (in minutes). This metric will be compared between conditions to evaluate the effect of the intervention.
Sleep macrostructure - Percentage of Time per Sleep Stage | Throughout Nights 1/2.
  Sleep macrostructure will be measured using the scoring manual of the American Academy of Sleep Medicine (AASM; Iber et al., 2007) as the established standard. Obtaining the sleep stage for each 30-sec epoch of the recording, allows calculating the percentage of time spent in each of the sleep stages: N1, N2, N3, REM, Wake (%). This metric will be compared between conditions to evaluate the effect of the intervention.
Sleep macrostructure - Sleep Efficiency | Throughout Nights 1/2.
  Sleep macrostructure will be measured using the scoring manual of the American Academy of Sleep Medicine (AASM; Iber et al., 2007) as the established standard. Obtaining the sleep stage for each 30-sec epoch of the recording, allows calculating the sleep efficiency (%), which represents the percentage of the night that is spent in actual sleep. This metric will be compared between conditions to evaluate the effect of the intervention.
Subjective sleep quality | Administered 0.5-1 hour before and after waking up on Nights 1 and 2.
  Subjective sleep quality will be measured using the SF-A-R questionnaire (German: "Schlaffragebogen A Revidierte Fassung"). This questionnaire measures 10 indices about sleep characteristics:
  * ESS (Difficulties falling asleep) -> 1-no difficulties / 5-very difficult
  * DSS (Difficulties staying asleep) -> 1-no difficulties / 5-very difficult
  * VZA (Early awakening) -> 1-did not wake up early / 5-woke too early
  * ASC (General sleep characteristics) -> 1-bad / 5-good sleep characteristics
  * GSD (Total sleep time) -> hours, minutes in decimal system
  * SQ (Sleep quality) -> 1-low / 5-high quality
  * GES (Feeling of recovery after sleep) -> 1-not recovered / 5-recovered
  * PSYA (Psychological balance before sleep) -> 1-imbalanced / 5-balanced
  * PSYE (Psychological exhaustion before sleep) -> 1-not exhausted / 5-exhausted
  * PSS (Psychosomatic symptoms during sleep) -> 1-none / 5-many
  These metrics will be compared between conditions to evaluate the effect of the intervention.
Subjective sleep quality | Administered 15 minutes before sleep onset and 15 minutes after waking up on Nights 1 and 2
  Sleepiness will be measured using the Stanford Sleepiness Scale. This test measures sleepiness in a range from 1 (wide awake) to 8 (fast asleep). This metric will be compared between conditions to evaluate the effect of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Bit&Brain Technologies SL, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes